CLINICAL TRIAL: NCT01451554
Title: Portion Control for the Treatment of Obesity in the Primary Care Setting
Brief Title: Portion Control Treatment for Obesity
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Jon Ebbert, Principal Investigator, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 02-003653
Record Dates: First submitted 2011-10-11; First posted 2011-10-13 (Estimated); Results first posted 2011-11-28 (Estimated); Last update posted 2011-11-28 (Estimated); Status verified 2011-10

CONDITIONS: Obesity
Keywords: weight; body mass index; obesity; portion control plate; diet; exercise
MeSH Terms: conditions — Obesity; Body Weight; Motor Activity | interventions — Nutrition Assessment

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Portion Control Intervention (Active Comparator): Individuals will be given a portion control plate and dietary counseling
  Interventions: Behavioral: portion control plate
- Usual Care (Placebo Comparator): Provided with self-help booklets on diet and exercise.
  Interventions: Behavioral: Usual Care

INTERVENTIONS:
Behavioral: portion control plate — Individuals are provided with a portion control plate to use while eating and dietary counseling by dietician
  Other Names: dietary counseling; weight loss intervention
  Arms: Portion Control Intervention
Behavioral: Usual Care — self-help booklets
  Other Names: self-help booklets(exercise and lifestyle changes)
  Arms: Usual Care

SUMMARY:
To date, no studies have been published assessing the effectiveness of portion control interventions in a primary care setting. The investigators will conduct a pilot study to assess the effectiveness of an intervention including a portion control plate and dietary counseling for weight loss among obese patients in a general medicine primary care practice.

DETAILED DESCRIPTION:
2-3 weeks prior to the patient's appointment with their primary care physician, the patient's medical record is reviewed to assess eligibility. If eligible, baseline patient characteristics are recorded, and a letter is sent to the patient informing them of the study and asking them to discuss this further with their primary care provider at their upcoming appointment.

At the primary care appointment, the patient is informed of the study and asked if they would like to participate. If the patient declines, their response is recorded. If the patient accepts, authorization is obtained and the patient is randomized by drawing a sealed envelope from either the male box or the female box, with both boxes being randomized. The envelope indicates either portion control plate or usual care. If the patient is randomized to usual care, Mayo Clinic pamphlets entitled "Lifestyle Changes for Healthy Weight" and "Exercise: Getting Started and Staying With It" are given to the patient. If the patient is randomized to the portion control plate, a 60 minute appointment with a dietician is scheduled. For pre-menopausal female patients who have not had a hysterectomy, a urine pregnancy test is performed to confirm that the patient is not pregnant prior to participation in the study.

At the dietitian appointment, the patient is given general information regarding portion size control and specific instructions on how to use a commercially calibrated portion control plate/bowl. The patient receives a handout containing instructions on how to use the plate/bowl along with food suggestions. The patient is instructed to use the plate for their largest meal of the day and encouraged to use the plate/bowl for all meals. The patient is also given a simple log-sheet to document the meals each day for which they used the plate/bowl.

The patients are then followed for 6 months. All patients are scheduled for weigh-ins at 3 months and 6 months. Patients in the portion control plate group are also contacted by phone or email (according to patient preference) at 1, 3, and 5 months by the dietitian to check-in and answer all questions. At completion of the study, patients in the portion control group are provided with a survey to assess their satisfaction with the intervention.

ELIGIBILITY:
Inclusion Criteria:

* Body Mass Index greater than 29 or less than 40
* Age between 18 and 75

Exclusion Criteria:

* Presence of active cancer
* Current participation in an organized weight loss program
* Current use of a weight loss medication
* History of bulimia or anorexia
* Current treatment for psychiatric illness other than anxiety or depression
* Surgery within the 3 months before enrollment or planned during the study period
* Past gastric bypass surgery or planned gastric bypass surgery during the - study period
* Current pregnancy or planned pregnancy during the study period

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2009-01; Primary Completion 2010-06 (Actual); Study Completion 2010-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jon O Ebbert, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

REFERENCES:
- [Result] Kesman RL, Ebbert JO, Harris KI, Schroeder DR. Portion control for the treatment of obesity in the primary care setting. BMC Res Notes. 2011 Sep 9;4:346. doi: 10.1186/1756-0500-4-346. PMID 21906302

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were referred to the study by their primary health care provider. Recruitment began on January 14, 2009 and ended on May 21, 2010.
Period: Overall Study
Arm/Group | Portion Control Intervention | Usual Care
Started | 33 | 32
Completed | 19 | 23
Not Completed | 14 | 9
Not completed — Withdrawal by Subject | 14 | 9

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Portion Control Intervention | Usual Care | Total
Number analyzed (Participants) | 33 | 32 | 65
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 28 | 24 | 52
  >=65 years | 5 | 8 | 13
Age Continuous [Mean (Standard Deviation); unit: years] | 55.4 (9.4) | 56.3 (10.7) | 55.9 (10.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 20 | 40
  Male | 13 | 12 | 25
Baseline Weight [Mean (Standard Deviation); unit: Kg] — Weight in Kilograms at the study entry
  Kg | 97.6 (12.8) | 98.8 (12.5) | 98.2 (12.6)

OUTCOME MEASURES:

1. Secondary Outcome: Weight Change at 3 Months
Description: Percentage change in weight at 3 months post study baseline
Time Frame: 3 months
Population: Intent to treat population includes all randomzied subjects. Missing data were imputed using the last observation carried forward.
Measure: Mean (Standard Deviation); unit: percentage
Arm/Group | Portion Control Intervention | Usual Care
Number analyzed (Participants) | 33 | 32
percentage | -1.7 (3.3) | -0.4 (1.9)
Statistical Analysis 1: Comparison: Portion Control Intervention vs Usual Care; Data were compared between groups using the 2 sample T-test; Test type: Superiority or Other; p = 0.06, t-test, 2 sided — 2 tailed t-test

2. Primary Outcome: Weight Change at 6 Months
Description: Weight change as a percentage of baseline at post 6 months.
Time Frame: 6 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage
Arm/Group | Portion Control Intervention | Usual Care
Number analyzed (Participants) | 33 | 32
percentage | -1.2 (3.1) | -0.4 (3.2)
Statistical Analysis 1: Comparison: Portion Control Intervention vs Usual Care; Data were compared between groups using a 2 sample T-test; Test type: Superiority or Other; p = 0.31, t-test, 2 sided

ADVERSE EVENTS:
Arm/Group | Portion Control Intervention | Usual Care
Serious Adverse Events (participants affected / at risk) | 0/33 | 0/32
Other Adverse Events (participants affected / at risk) | 0/33 | 0/32

LIMITATIONS AND CAVEATS:
small sample size and inability to blind staff/study subject to the intervenion

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes